CLINICAL TRIAL: NCT02306577
Title: STRIBILD in Non-Nucleoside Resistant Patients, An Evaluation of Safety and Efficacy in Vulnerable Population (SINNR STUDY)
Brief Title: STRIBILD in Non-Nucleoside Resistant Patients (SINNR STUDY)
Acronym: SINNR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vancouver Infectious Diseases Centre (Other)
Collaborators: Gilead Sciences (Industry); Regina General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SINNR STUDY
Record Dates: First submitted 2014-11-05; First posted 2014-12-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: HIV; Illicit Drug User
Keywords: STRIBILD; HIV; Illicit dgug user
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vancouver: HIV infected people who are current of recent illicit drug users and receive Stribild for their HIV treatment at Vancouver Infectious Diseases Centre and Regina General Hospital.
  Interventions: Drug: STRIBILD

INTERVENTIONS:
Drug: STRIBILD — Taking oral 1 STRIBILD tablet once a day for 48 weeks

SUMMARY:
The SINNR study will evaluate the virologic efficacy (viral load <50 copies/mL)and safety of STRIBILD administered for 48 weeks to HIV-infected current or recent illicit drug users.

DETAILED DESCRIPTION:
The SINNR study is a pilot, observational, open label study. It will evaluate the virologic efficacy (viral load <50 copies/mL), safety, and immunologic response of STRIBILD administered for 48 weeks to HIV-infected current or recent illicit drug users.

Approximately 30 HIV-infected current or recent illicit drug users (≥19y.o.,<70y.o.) from Vancouver Infectious Diseases Centre and Regina General Hospital, University of Saskatchewan will be taking an oral 1 STRIBILD tablet once a day for 48 weeks.

Additionally, adherence to STRIBILD over 48 weeks and quality of life will be measured in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is at least 19 years of age and less than 70 years of age infected with HIV and requiring antiretroviral therapy on medical grounds and who has acquired HIV infection through illicit drug use.
2. Participant has documented resistance to NNRTIs, with the presence of one or more primary resistance mutations (Stanford database), on current or previous therapy.
3. The primary care provider decides to prescribe STRIBILD.
4. Participant has no ongoing issues that would lead to significant non-compliance with the study procedures even in the presence of optimal adherence support structures.
5. Participant is able to read and write in the language of the questionnaires and give informed consent.
6. Participant must not be taking any medication that could interact with STRIBILD.
7. If female, participant must have a negative pregnancy test and agree to use, for the duration of the study, a method of birth control that has a history of proven reliability as judged by the investigator.

Exclusion Criteria:

1. Participant has previous exposure to STRIBILD.
2. Participant has documented resistance to any of the components of STRIBILD.
3. Participant is pregnant or breast-feeding.
4. Participant has a contraindication to the use of STRIBILD for any reason.
5. Participant has active hepatitis B (HbsAg positive).
6. Participant has any of the following abnormal laboratory test results at screening:

   Hemoglobin less than 10.0 g/dL, Absolute neutrophil count less than 750 cells/mL, Platelet count less than 50,000/mL, ALT or AST less than 5x Upper Limit of Normal (ULN), Creatinine less than 1.5 x ULN.
7. Participant, in the opinion of the principal investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected people who are current or past illicit drug users and receive treatment for their HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Virologic Efficacy (viral load <50copies/ml after taking STRIBILD) | 48 weeks
  Evaluate viral load <50copies/ml after taking STRIBILD

SECONDARY OUTCOMES:
Safety-Side Effect Profile and Number of Participants with Adverse Events | 48 weeks
  Evaluate safety of STRIBILD
Immunologic Response-CD4 Cell Count and Change in CD4 Cell Count at 48 Weeks | 48 weeks
  Evaluate immunologic response of STRIBILD
Adherence | 48 weeks
  Evaluate Adherence to STRIBILD
Quality of Life | 48 weeks
  Evaluate Quality of life after taking STRIBILD

CONTACTS AND LOCATIONS:
Overall Officials: Brian Conway, MD, Principal Investigator — Vancouver ID Research and Care Centre Society
Locations (1):
- Vancouver ID Research and Care Centre Society, Vancouver, British Columbia, Canada